CLINICAL TRIAL: NCT02033707
Title: Phase I Study Characterizing Effects of Hallucinogens and Other Drugs on Mood and Performance
Brief Title: Effects of Hallucinogens and Other Drugs on Mood and Performance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NA_00082804
Record Dates: First submitted 2013-12-30; First posted 2014-01-13 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Healthy
Keywords: Hallucinogen; Cognitive effects; Subjective effects
MeSH Terms: interventions — Hallucinogens; Hypnotics and Sedatives; Anti-Anxiety Agents; Histamine Antagonists; Central Nervous System Stimulants; Analgesics, Opioid; Ethanol; Scopolamine; Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Male volunteers (Experimental): Hallucinogens and psychoactive substances will be administered via capsule. Results will be compared between male and female participants.
  Interventions: Drug: Hallucinogens and psychoactive substances
- Female volunteers (Experimental): Hallucinogens and psychoactive substances will be administered via capsule. Results will be compared between male and female participants.
  Interventions: Drug: Hallucinogens and psychoactive substances

INTERVENTIONS:
Drug: Hallucinogens and psychoactive substances — One of the following or placebo will be given:
  Hallucinogens: DMT, 4-phosphoryloloxy-N-diethyltryptamine, dipropyltryptamine (DPT), ketamine, dextromethorphan, mescaline, PCP, psilocybin, salvinorin-A, LSD, d-lysergic acid amide (LSA), MDMA, cannabis
  Sedatives/anxiolytics: alprazolam, diazepam, lorazepam, secobarbital, temazepam, triazolam, zolpidem
  Antihistamines: diphenhydramine, chlorpheniramine
  Stimulants: d-amphetamine, caffeine, ephedrine, methylphenidate, diethylproprion
  Opioids: heroin, morphine, oxycodone, hydrocodone, methadone, codeine
  Other: alcohol, scopolamine, nicotine
  Each volunteer will receive a hallucinogen on at least one of five sessions. More drugs are listed than will be administered to increase the degree to which volunteers are "blind" to the drugs being studied. It is important that the volunteer and research staff be blinded to specific drug conditions to minimize confounding the results with expectations about the nature of drug effects.
  Other Names: Hallucinogens; Sedatives & anxiolytics; Antihistamines; Stimulants; Opioids; Alcohol; Scopolamine; Nicotine

SUMMARY:
This non-treatment study will investigate the effects on mood and performance caused by hallucinogens and other psychoactive compounds.

DETAILED DESCRIPTION:
Twenty volunteers between 21-50 years old will each participate in 16 total sessions, including sessions for: screening, preparation, experiment/drug, immediate follow-ups, a 1-month follow-up and 1 post completion urine collection. On each of five experimental session participants will orally ingest capsules of either a placebo or varying doses of one of 18 different psychoactive compounds.

Subjective drug effects will be examined with methods previously used by this laboratory for characterizing the effects of psychoactive substances from a variety different classes. Volunteers will swallow capsules containing various doses of drugs, complete tasks during the session, and rate effects of the drug and complete questionnaires at the end of each session as described below.

ELIGIBILITY:
Inclusion Criteria:

* Be 21 to 50 years old
* Have given written informed consent
* Have a high school level of education
* Have a self-reported interest in psychedelic drugs and altered states of consciousness
* Have used classic, serotonergic hallucinogens or dissociative anesthetic hallucinogens (e.g., LSD, psilocybin mushrooms, ayahuasca, ketamine, PCP) without untoward effects. Volunteers must report "liking" of psychedelic and psychedelic-like drugs and report having used hallucinogens at least 5 times in their lifetime and at least once within the last 2 years
* Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the mornings of drug session days. If the volunteer does not usually consume caffeinated beverages, he or she must agree not to do so on session days
* Cigarette smokers must agree to abstain from smoking on session days from 1 hour before drug administration until at least 6 hours after drug administration
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages, within 24 hours of each drug administration. Exceptions include daily use of caffeine and nicotine.
* Be healthy and psychologically stable as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests
* Agree that for one week before each session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the study investigators. Exceptions will be evaluated by the study investigators and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals
* Agree not to take any PRN prescription medications on the mornings of the sessions
* Be willing and able to participate

Exclusion criteria:

* Women who are pregnant (as indicated by a positive urine pregnancy test assessed at intake and before each drug session) or nursing; women who are of child-bearing potential and sexually active who are not practicing an effective means of birth control
* Cardiovascular conditions: coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant ECG abnormality (e.g., atrial fibrillation), or TIA in the past year
* Epilepsy with history of seizures
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* Currently taking psychoactive prescription medication on a regular (e.g., daily) basis
* Currently taking on a regular (e.g., daily) basis any medications having a primary centrally-acting pharmacological effect on serotonin neurons or medications that are MAO inhibitors. For individuals who have intermittent or PRN use of such medications, sessions will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose
* More than 20% outside the upper or lower range of ideal body weight

Psychiatric Exclusion Criteria:

* Current or past history of meeting DSM-IV criteria for schizophrenia, psychotic disorder (unless substance-induced or due to a medical condition), or bipolar I or II disorder
* Current severe obsessive-compulsive disorder, dysthymic disorder, or panic disorder.
* Current, severe, major depression
* Have a first or second degree relative with schizophrenia, psychotic disorder (unless substance induced or due to a medical condition), or bipolar I or II disorder
* Currently meets DSM-IV criteria for dissociative disorder, anorexia nervosa, bulimia nervosa, or other psychiatric conditions judged to be incompatible with establishment of rapport or safe exposure to study compounds

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Rating of "Drug Liking" on the End of Day Questionnaire | Completed at the end of the experimental session (approximately 8 hours after capsule administration)
  Volunteer-completed questionnaire assesses the subjective liking of the drug condition for the session

SECONDARY OUTCOMES:
Hallucinogen Rating Scale | Completed at the end of the experimental session (approximately 8 hours after capsule administration)
  This questionnaire has been used in various studies to characterize the profile of subjective and cognitive effects of various types of drugs classified as hallucinogens

CONTACTS AND LOCATIONS:
Overall Officials: Roland R Griffiths, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Mathai DS, Hilbert S, Sepeda ND, Strickland JC, Griffiths RR, Garcia-Romeu A. Double-Blind Comparison of the Two Hallucinogens Dextromethorphan and Psilocybin: Experience-Dependent and Enduring Psychological Effects in Healthy Volunteers. Psychedelic Med (New Rochelle). 2023 Dec 1;1(4):241-252. doi: 10.1089/psymed.2023.0035. Epub 2023 Dec 13. PMID 38152462